CLINICAL TRIAL: NCT00977808
Title: Pilot Study of Closed-Loop Glucose Control in People With Type 1 Diabetes(BPK004)
Brief Title: Pilot Study of Closed-Loop Glucose Control in People With Type 1 Diabetes (BPK004)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Boris Kovatchev, PhD, Professor, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12998; BPK004
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Type 1 Diabetes
Keywords: Artificial pancreas; Closed-Loop control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-Loop Model Predictive Control (MPC) (Experimental): Insulin dosing was performed by a model-predictive control (MPC) algorithm.
  Interventions: Device: Closed-Loop, Model Predictive Control (MPC)
- Open-Loop (Placebo Comparator): Insulin dosing was performed by the patient (using their normal routine and personal insulin pump) under a physician's supervision.
  Interventions: Device: Open-Loop

INTERVENTIONS:
Device: Closed-Loop, Model Predictive Control (MPC) — Subjects used the OmniPod Insulin Management System (Insulet Corp.) and Insulin lispro (Eli Lilly, Indianapolis, IN). MPC algorithm suggested insulin boluses every 15 min, which, if accepted, were programmed into the insulin pump by the attending physician. Otherwise, the admission remained the same as in the open-loop admission (i.e. meals, sleep, etc...).
  Arms: Closed-Loop Model Predictive Control (MPC)
Device: Open-Loop — This admission was to assess the subjects' level of glucose control and created a base to compare the performance of the closed-loop system. Subjects monitored their own blood glucose values and administer their basal/bolus as they would at home. Subjects used their own insulin pumps and Insulin lispro (Eli Lilly, Indianapolis, IN). Otherwise, the admission remained the same as in the closed-loop admission (i.e. meals, sleep, etc...).
  Arms: Open-Loop

SUMMARY:
This study plans to link two existing technologies, the insulin pump and the continuous glucose monitor (CGM), to essentially develop an artificial pancreas, i.e., closed-loop. This will be done using two continuous glucose monitors (CGMs), a computer containing an investigational control algorithm that uses glucose information from the CGM to recommend insulin dosing, and an insulin pump. The purpose of this study is to test the ability of continuous glucose monitors together with an insulin pump and a mathematical formula to control blood sugar levels of people with type 1 diabetes.

The Closed-Loop control algorithm will:

1. Suggest adequate insulin delivery for blood glucose control in steady state (overnight);
2. Cover adequately with an insulin bolus the pre-set carbohydrate content of a breakfast.

If successful, this study will conceptually prove the feasibility of automated model-predictive closed-loop glucose control in T1DM.

DETAILED DESCRIPTION:
Each patient had an outpatient screening evaluation, and two 22 h overnight hospital admissions separated by a 2- to 4-week waiting period. Each inpatient admission began at 15:00 and ended at 13:00 on the following day. Subjects ate dinners and lunches with carbohydrate content that was the same at admission 1 and admission 2 and had identical morning meals of Ensure Plus (Abbott Nutrition, Columbus, OH). Two days before each admission, two Freestyle Navigator CGM devices (Abbott Diabetes Care) continuous glucose monitors were applied to the patient to allow for stabilization of the sensors and for assessment of their performance.

During admission 1, open-loop control was used, with the subjects' usual insulin routine and their personal insulin pump. During admission 2, an OmniPod Insulin Management System (Insulet Corp.) was inserted and used for closed-loop control of blood glucose. Insulin lispro (Eli Lilly, Indianapolis, IN), chosen based on commercial assays available, was used during both inpatient admissions.

At the beginning of admission 2, one of the two CGM devices was designated as primary, and the closed-loop control algorithm used the data of that system, unless a problem was detected. At 17:00, the model-predictive control (MPC) was initiated in a data-collection mode, automatically receiving CGM data every minute. Administration of the predinner insulin bolus was overseen by the attending physician. MPC, closed-loop control began at 21:30 and continued until 12:00 the next day for a total of 14.5 h.

Per FDA restrictions, the algorithm did not automatically control the insulin pump. Instead, the algorithm suggested insulin boluses every 15 min, which, if accepted, were programmed into the insulin pump by the attending physician. This was done for safety reasons, allowing the physician to override insulin delivery suggestions at any time. Reference blood glucose (using a YSI Life Sciences or a Beckman glucose analyzer) was sampled every 30 min. The protocol required switching to more frequent 15 min reference blood glucose sampling if hypoglycemia occurred or was imminent. Fast-acting carbohydrate (glucose tablets or fruit juice) was given when reference blood glucose fell below 3.9 mmol/liter, regardless of the CGM readings.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Have Type 1 Diabetes Mellitus as defined by American Diabetes Association criteria or judgment of physician for at least 2 years (including those who may also be treated with metformin, thiazolidinedione, exenatide, or pramlintide).
* Use of an insulin pump
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 1 month prior to enrollment in the study
* Willingness to use lispro (Humalog) insulin for the duration of the inpatient study
* Demonstration of proper mental status and cognition for the study

Exclusion Criteria:

* Age <21
* Pregnancy
* Hematocrit <36% (females); <38% (males)
* Symptomatic coronary artery disease (e.g. history of myocardial infarction, history of acute coronary syndrome, history of therapeutic coronary intervention, history of coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, positive stress test or catheterization with coronary blockages >50%).
* Congestive heart failure
* History of a cerebrovascular event
* Use of a medication that significantly impacts glucose metabolism (oral steroids)
* Atrial fibrillation
* Uncontrolled hypertension (resting blood pressure >140/90)
* History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans
* Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the FreeStyle NavigatorTM CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
* Active enrollment in another clinical trial
* Allergy or adverse reaction to lispro insulin
* Known adrenal gland problem, pancreatic tumor, or insulinoma
* Current alcohol abuse, substance abuse, or severe mental illness
* Retinopathy and renal failure
* Uncontrolled anxiety or panic disorder
* Known bleeding diathesis or dyscrasia
* Renal insufficiency (creatinine >1.5)
* Any comorbid condition affecting glucose metabolism

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris P Kovatchev, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Kovatchev B, Cobelli C, Renard E, Anderson S, Breton M, Patek S, Clarke W, Bruttomesso D, Maran A, Costa S, Avogaro A, Dalla Man C, Facchinetti A, Magni L, De Nicolao G, Place J, Farret A. Multinational study of subcutaneous model-predictive closed-loop control in type 1 diabetes mellitus: summary of the results. J Diabetes Sci Technol. 2010 Nov 1;4(6):1374-81. doi: 10.1177/193229681000400611. PMID 21129332

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults With Type 1 Diabetes: During admission 1, open-loop control was used, with the subjects' usual insulin routine and their personal insulin pump.
  At the beginning of admission 2 (closed-loop control), one of the two CGM devices was designated as primary, and the closed-loop control algorithm used the data of that system, unless a problem was detected. At 17:00, the model-predictive control (MPC) was initiated in a data-collection mode, automatically receiving CGM data every minute. Administration of the predinner insulin bolus was overseen by the attending physician. MPC, closed-loop control began at 21:30 and continued until 12:00 the next day for a total of 14.5 h. Per FDA restrictions, the algorithm did not automatically control the insulin pump. Instead, the algorithm suggested insulin boluses every 15 min, which, if accepted, were programmed into the insulin pump by the attending physician.
Period: Overall Study
Arm/Group | Adults With Type 1 Diabetes
Started | 12
Completion of Open-Loop Admission | 12
Completion of Closed-Loop Admission | 11
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adults With Type 1 Diabetes
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.17 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Hypoglycemic Episodes
Description: Hypoglycemic events were defined as below 3.9 mmol/liter and the percentage of time within the range of 3.9 to 7.8 mmol/liter overnight (21:30 until 08:00) as measured by reference blood glucose (YSI or Beckman Glucose Analyzer).
Time Frame: Overnight (21:30 until 08:00)
Population: Only participants who completed both study periods were considered for this assessment.
Measure: Number; unit: Hypoglycemic Episodes
Groups:
- Experimental: Closed-Loop Model Predictive Control (MPC): Insulin dosing was performed by a model-predictive control (MPC) algorithm.
- Control: Open-Loop: Insulin dosing was performed by the patient (using their normal routine and personal insulin pump) under a physician's supervision.
Arm/Group | Experimental: Closed-Loop Model Predictive Control (MPC) | Control: Open-Loop
Number analyzed (Participants) | 11 | 11
Hypoglycemic Episodes | 5 | 23

ADVERSE EVENTS:
Arm/Group | Adults With Type 1 Diabetes
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes